CLINICAL TRIAL: NCT00787761
Title: Pre-administration of Rabbit Antithymocyte Globulin to Optimize Donor T-Cell Engraftment Following Reduced Intensity Allogeneic Peripheral Blood Progenitor Cell Transplantation From Matched-Related Donors
Brief Title: Early Administration of ATG Followed by Cyclophosphamide, Busulfan and Fludarabine Before a Donor Stem Cell Transplant in Patients With Hematological Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000618483; BMTGG-NSH-807
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-08

CONDITIONS: Myeloproliferative Disorders; Kidney Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: accelerated phase CML; blastic phase CML; Philadelphia chromosome positive CML; stage I CLL; stage II CLL; stage III CLL; stage IV CLL; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; adult AML with 11q23 (MLL) abnormalities; adult CML in remission; adult ALL in remission; stage IV renal cell cancer; de novo MDS; previously treated MDS; secondary MDS; atypical CML, BCR-ABL negative; chronic myelomonocytic leukemia; MDS/myeloproliferative neoplasm, unclassifiable; primary myelofibrosis; chronic neutrophilic leukemia; recurrent adult Hodgkin lymphoma; clear cell renal cell carcinoma; adult AML with inv(16)(p13;q22); adult AML with t(15;17)(q22;q12); adult AML with t(16;16)(p13;q22); adult AML with t(8;21)(q22;q22); adult nasal type extranodal NK/T-cell lymphoma; AML/transient myeloproliferative disorder; Burkitt lymphoma; chronic phase CML; extranodal marginal zone B-cell lymphoma of mucosa tissue; nodal marginal zone B-cell lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; recurrent adult diffuse mixed cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; contiguous st II adult diffuse small cleaved cell lymphoma; noncontiguous st II diffuse small cleaved cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; recurrent adult grade III lymphomatoid granulomatosis; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; splenic marginal zone lymphoma; Waldenstrom macroglobulinemia; recurrent adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Kidney Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Congenital Abnormalities; Carcinoma, Renal Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Hodgkin Disease; Leukemia, Promyelocytic, Acute; Lymphoma, Extranodal NK-T-Cell; Burkitt Lymphoma; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; Cyclophosphamide; fludarabine phosphate; Methotrexate; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATG, Cytoxan, Bu/Flu based Allogeneic Transplant (Experimental): All patients will receive an ATG, Cyclosphosphamide, Busulfan and Fludarabine based Allogeneic Transplant
  Interventions: Biological: anti-thymocyte globulin; Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methotrexate; Drug: tacrolimus; Procedure: nonmyeloablative allogeneic HSCT

INTERVENTIONS:
Biological: anti-thymocyte globulin — Anti-Thymocyte Globulin (ATG) is commercially available. The 1st vial contains 25 mg ATG, and the 2nd vial contains > 5 mL SWFI diluent. Ampuls must be refrigerated (2º C - 8º C). Do not freeze.
  Reconstitute 25 mg vial with diluent provided by manufacturer. Roll vial gently to dissolve powder. Use contents of vial within 4 hours. Dilute dosage to a final concentration of 0.5 mg/mL in 0.9% sodium chloride injection or 5% dextrose injection. Gently invert admixture 1-2 times to mix. Use admixture solution immediately.
  Infuse the 1st dose over at least 6 hours, and subsequent doses over at least 4 hours. Infuse through a 0.22 micron in-line filter. Premeds include acetaminophen 650 mg PO, diphenhydramine 25-50 mg PO/IV, and methyprednisolone 1mg/kg at the initiation and half-way through ATG administration.
  Other Names: Thymoglobulin; ATG
Drug: busulfan — Commercially available in 60 mg/10 mL ampuls.
  Dilute busulfan injection in 0.9% sodium chloride injection or dextrose 5% in water. The dilution volume should be 10 times the volume of busulfan injection, ensuring that the final concentration of busulfan is ≥ 0.5 mg/mL.
  Store unopened ampuls at 2º C to 8º C. The diluted solution is stable for up to 8 hours at room temperature (25º C) but the infusion must also be completed within that 8-hour time frame. Dilution of busulfan injection in 0.9% sodium chloride is stable for up to 12 hours under refrigeration (2º C to 8º C) but the infusion must also be completed within that 12-hour time frame.
  IV Bu should be administered via a central venous catheter as a 2-hour infusion every 6 hours for 2 consecutive days for a total of 8 doses.
Drug: cyclophosphamide — Cyclophosphamide is commercially available. Cyclophosphamide for injection is available in 2000 mg vials which are reconstituted with 100 ml sterile water for injection.
  The concentration of the reconstituted product is 20 mg/ml. The calculated dose will be diluted further in 250-500 ml of Dextrose 5% in water.
  Reconstituted solutions of lyophilized cyclophosphamide are chemically and physically stable for 24 hours at room temperature or for 6 days in the refrigerator. Specific temperatures are not provided by the manufacturer. Reconstitution of cyclophosphamide with bacteriostatic water containing benzyl alcohol preservative may result in decomposition.
  Each dose will be infused over 1-2 hr (depending on the total volume).
Drug: fludarabine phosphate — Fludarabine is commercially available as a white, lyophilized powder. Each vial contains 50 mg of fludarabine, 50 mg of mannitol and sodium hydroxide to adjust pH.
  Intact vials should be stored under refrigeration. Reconstituted vials are stable for 16 days and solutions diluted in D5W or NS are stable for 48 hours at room temperature or under refrigeration.
  Fludarabine should be reconstituted with 2 mL of Sterile Water for Injection, USP. Each mL of the resulting solution will contain 25 mg of fludarabine, 25 mg of mannitol, and sodium hydroxide to adjust the pH to 7-8.5. The product should be further diluted for intravenous administration in 5% Dextrose for Injection, USP or in 0.9% Sodium Chloride, USP.
  Fludarabine will be administered as an IV infusion over 30 minutes.
  Other Names: Fludara
Drug: methotrexate — Commercially available for injection in 2 mL (2.5 mg/mL), 2 mL, 4 mL, 8 mL, 10 mL (25 mg/mL) vials, or 20 mg, 25 mg, 50 mg, or 100 mg vials for reconstitution.
  Vials requiring reconstitution should be reconstituted to a concentration of 25 mg/mL.
  Intact vials should be stored at room temperature and protected from light. Once opened, solutions containing preservatives are stable for 4 weeks at room temperature and up to 3 months refrigerated.
  Administer via slow IV push.
  Other Names: Amethopterin, MTX
Drug: tacrolimus — Tacrolimus is commercially available as an injection (5 mg/mL; 1 mL ampuls) and as oral capsules (1 mg and 5 mg).
  Tacrolimus injection must be diluted prior to IV infusion with 0.9% sodium chloride or 5% dextrose injection to a concentration of 4-20 μg/mL. Solutions should be prepared in non-PVC plastic or glass. Tacrolimus injection and diluted solutions of the drug should be inspected visually for particulate matter and discoloration prior to administration whenever solution and container permit.
  Oral therapy should be started as possible as per protocol and 8 to 12 hours after stopping intravenous therapy. Oral doses will be administered twice a day.
  Store tacrolimus capsules and injection at controlled room temperature, 15-30º C (59-86º F).
  Other Names: Prograf, FK506
Procedure: nonmyeloablative allogeneic HSCT — As demonstrated by groups in Houston, Jerusalem & Seattle, RICT has been used to treat hematologic & solid malignancies with related & unrelated donors. Although adequate comparisons of RICT versus ablative alloHCT remain to be reported, the studies of RICT so far suggest that TRM is generally less than would be expected for similar patients undergoing ablative alloHCT; incidence of acute & chronic GVHD is similar or less than ablative alloHCT; autologous hematopoietic recovery is more common than seen following ablative alloHCT if graft failure occurs; powerful GVT effects can be seen but are dependent on high levels of donor T-cell chimerism and RICT are less effective than ablative alloHCT in controlling aggressive malignancies

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving antithymocyte globulin before the transplant and tacrolimus and methotrexate after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving antithymocyte globulin together with cyclophosphamide, busulfan, and fludarabine works in treating patients with hematological cancer or kidney cancer undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the percentage of patients with hematological malignancies or renal cell carcinoma who achieve > 90% donor T-cell chimerism at 30 days after treatment with reduced-intensity conditioning comprising low-dose anti-thymocyte globulin, low-dose cyclophosphamide, busulfan, and fludarabine phosphate followed by allogeneic peripheral blood progenitor cell transplantation from a matched related donor.
* To assess the incidence of severe (grade 3 or 4) acute graft-versus-host disease (GVHD) and extensive chronic GVHD in these patients.
* To assess whether this regimen is associated with reduced transplant-related toxicity and increased tolerability in these patients.
* To assess the overall safety of this conditioning regimen as measured by 6-month transplant-related mortality in these patients.
* To determine the efficacy of this regimen in inducing durable remissions in these patients.

OUTLINE:

* Reduced-intensity conditioning (RIC): Patients receive anti-thymocyte globulin IV over 4-6 hours on day -16 and over 6-8 hours on day -15, fludarabine phosphate IV over 30 minutes on days -7 to -3, busulfan IV over 3 hours on days -4 and -3, and cyclophosphamide IV over 1-2 hours on day -2.
* Transplantation: Patients undergo allogeneic peripheral blood progenitor cell transplantation on day 0.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive oral tacrolimus every 12 hours on days -1 to 90, followed by a taper until day 150. Patients also receive methotrexate IV on days 1, 3, and 6.

Blood samples are collected periodically for pharmacokinetic studies of anti-thymocyte globulin and PCR analysis for chimerism.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one of the following:

  * Chronic myeloid leukemia (CML)

    * Philadelphia chromosome (Ph)- and/or BCR-ABL-positive disease
    * In chronic or accelerated phase
    * Suboptimal response to imatinib mesylate (i.e., no hematologic complete response by 3 months, no major cytogenetic response by 6 months, or no complete cytogenetic response by 1 year)
    * CML in blastic transformation allowed provided patient achieved complete remission (CR) or second chronic phase after treatment with imatinib mesylate or chemotherapy
  * Chronic lymphocytic leukemia meeting one of the following criteria:

    * Rai stage III or IV disease
    * Rai stage I or II disease that failed standard therapy (i.e., disease is progressing after ≥ 1 course of standard therapy)
  * Non-Hodgkin lymphoma (NHL) meeting one of the following criteria:

    * Indolent NHL

      * Clinical stage III or IV disease or bulky stage II disease (i.e., ≥ one lymphoid mass > 5 cm in ≥ one dimension)
      * Relapsed after primary therapy OR is refractory to therapy
    * Aggressive NHL

      * Is not considered curable with standard chemotherapy or autologous stem cell transplantation (i.e., relapsed after autologous stem cell transplantation)
      * Chemotherapy-responsive disease
  * Multiple myeloma

    * Durie-Salmon stage II or III disease

      * Durie Salmon stage I disease allowed provided β2 microglobulin level > 3 mg/dL
  * Acute myeloid leukemia or acute lymphocytic leukemia

    * In CR (defined as < 5% blasts in bone marrow and no circulating blasts) AND has any of the following poor prognostic features:

      * WBC > 100,000/mm^3 at presentation
      * In second or greater remission
      * Adverse-risk cytogenetics (i.e., Ph1-positive, 11q23 translocation, -5, -7, complex translocations, or other recognized adverse-risk cytogenetics)
  * Renal cell carcinoma

    * Stage IV disease
    * Clear cell morphology
  * Myelodysplastic syndromes

    * Bone marrow blasts ≤ 10% on last bone marrow biopsy prior to transplantation
  * Myeloproliferative disease

    * Anticipated life expectancy on conventional therapy < 10 years
    * No uncomplicated essential thrombocythemia or primary polycythemia
  * Hodgkin lymphoma

    * Relapsed after ≥ 1 standard-dose chemotherapy regimen
    * Not considered curable by autologous stem cell transplantation
* No clinical evidence of active CNS involvement

  * Previously treated leptomeningeal disease allowed provided CSF cytology is negative at the time of assessment for transplantation
* Available 6/6 allele match (i.e., HLA-A, B, DRβ1)matched related donor

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Bilirubin < 3 times normal (unless abnormality due to malignancy)
* AST and ALT < 3 times normal (unless abnormality due to malignancy)
* Creatinine ≤ 2.0 mg/dL
* LVEF ≥ 40% by MUGA or ECHO
* DLCO ≥ 40% of predicted
* FEV-1 ≥ 50% of predicted
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Deemed to be an appropriate candidate for allogeneic SCT
* No evidence of myocardial infarction within the past 6 months
* No psychological or social condition that may interfere with study participation
* No serious uncontrolled localized or active systemic infection
* No second malignancy within the past 3 years except for completely excised nonmelanotic skin cancer or in situ carcinoma of the cervix
* No chronic inflammatory disorder requiring the continued use of glucocorticoids or other immunosuppressive medications
* No known HIV positivity
* No hypersensitivity to E. coli-derived proteins

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2010-07 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asad Bashey, MD, PhD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia, United States

REFERENCES:
- [Background] Rao SS, Peters SO, Crittenden RB, Stewart FM, Ramshaw HS, Quesenberry PJ. Stem cell transplantation in the normal nonmyeloablated host: relationship between cell dose, schedule, and engraftment. Exp Hematol. 1997 Feb;25(2):114-21. PMID 9015211
- [Background] Storb R, Yu C, Wagner JL, Deeg HJ, Nash RA, Kiem HP, Leisenring W, Shulman H. Stable mixed hematopoietic chimerism in DLA-identical littermate dogs given sublethal total body irradiation before and pharmacological immunosuppression after marrow transplantation. Blood. 1997 Apr 15;89(8):3048-54. PMID 9108426
- [Background] Giralt S, Estey E, Albitar M, van Besien K, Rondon G, Anderlini P, O'Brien S, Khouri I, Gajewski J, Mehra R, Claxton D, Andersson B, Beran M, Przepiorka D, Koller C, Kornblau S, Korbling M, Keating M, Kantarjian H, Champlin R. Engraftment of allogeneic hematopoietic progenitor cells with purine analog-containing chemotherapy: harnessing graft-versus-leukemia without myeloablative therapy. Blood. 1997 Jun 15;89(12):4531-6. PMID 9192777
- [Background] Slavin S, Nagler A, Naparstek E, Kapelushnik Y, Aker M, Cividalli G, Varadi G, Kirschbaum M, Ackerstein A, Samuel S, Amar A, Brautbar C, Ben-Tal O, Eldor A, Or R. Nonmyeloablative stem cell transplantation and cell therapy as an alternative to conventional bone marrow transplantation with lethal cytoreduction for the treatment of malignant and nonmalignant hematologic diseases. Blood. 1998 Feb 1;91(3):756-63. PMID 9446633
- [Background] McSweeney PA, Niederwieser D, Shizuru JA, Sandmaier BM, Molina AJ, Maloney DG, Chauncey TR, Gooley TA, Hegenbart U, Nash RA, Radich J, Wagner JL, Minor S, Appelbaum FR, Bensinger WI, Bryant E, Flowers ME, Georges GE, Grumet FC, Kiem HP, Torok-Storb B, Yu C, Blume KG, Storb RF. Hematopoietic cell transplantation in older patients with hematologic malignancies: replacing high-dose cytotoxic therapy with graft-versus-tumor effects. Blood. 2001 Jun 1;97(11):3390-400. doi: 10.1182/blood.v97.11.3390. PMID 11369628
- [Background] Champlin R, Khouri I, Anderlini P, De Lima M, Hosing C, McMannis J, Molldrem J, Ueno N, Giralt S. Nonmyeloablative preparative regimens for allogeneic hematopoietic transplantation. Biology and current indications. Oncology (Williston Park). 2003 Jan;17(1):94-100; discussion 103-7. PMID 12599934
- [Background] Platzbecker U, Ehninger G, Schmitz N, Bornhauser M. Reduced-intensity conditioning followed by allogeneic hematopoietic cell transplantation in myeloid diseases. Ann Hematol. 2003 Aug;82(8):463-468. doi: 10.1007/s00277-003-0680-7. Epub 2003 Jun 21. PMID 12910373
- [Background] Storb R. Non-myeloablative allogeneic transplantation -- state-of-the-art. Pediatr Transplant. 2004 Jun;8 Suppl 5:12-8. doi: 10.1111/j.1398-2265.2004.00189.x. PMID 15125701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 patients were enrolled between 4/20/2007 and 5/3/2010. Patients who were undergoing transplant at Northside Hospital were potentially eligible.
Pre-assignment Details: 29 patients signed consent for this study. 2 patients were initially screen failures but eventually were determined eligible & were treated on study. 1 patient was considered a screen failure due to having an ineligible donor. One patient had progressive disease and one patient had compliance-related issues prohibiting them from particiapting.
Groups:
- RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan: All patients received ATG 1mg/kg Day-16 and then 3.5 mg/kg Day -15 Fludarabine 30mg/m2/day on days -7 to -3 Busulfan 130 mg/m2 on days -4 & -3 Cyclophosphamide 1.5 g/m2 on day -2 Tacrolimus begins 0.03mg/kg bid on Day -1 Stem Cell transplant on Day 0 Methotrexate 5mg/m2 given D+1, +3 and +6
Period: Overall Study
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Achievement of > 90% (Full) Donor Chimerism in the T-cell Lineage as Measured by PCR at Day 30 Post-transplantation
Description: Chimerism analysis of peripheral blood mononuclear cells using PCR for STR/VNTR will be performed post transplant. On each occasion, the peripheral blood will be separated into the T-cell component (using e.g. CD3 selection) and the myeloid component (using e.g.CD14/15 selection) before assessment of chimerism.
Time Frame: Day 30
Population: only 15 of the patients treated on study had Day 30 chimerism results.
Measure: Number; unit: participants
Groups:
- Transplant Recipients: patients receiving transplant using ATG/Bu/Flu/Cy per this protocol
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 15
participants | 12

2. Secondary Outcome: T-cell and Myeloid Chimerism at Days 90 Post-transplantation (>90% Chimerism)
Description: as for outcome 1
Time Frame: Day 90
Population: 20 of the patients treated on this study had Day 90 chimerism drawn.
Measure: Number; unit: participants
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Number analyzed (Participants) | 20
participants | 17

3. Secondary Outcome: T-cell and Myeloid Chimerism at Days 180 Post-transplantation (>90%)
Description: as for outcome 1
Time Frame: 180 days
Population: 20 of the patients treated on study had chimerism drawn on day 180.
Measure: Number; unit: participants
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Number analyzed (Participants) | 20
participants | 19

4. Secondary Outcome: Number of Patients Who Experience Severe (Grade 3 or 4) Acute Graft-versus-host Disease
Description: number of patients who experienced post-transplant complication (GVHD) as seen by clinical evidence including but not limited to skin rash, elevated liver function tests, nausea/vomiting/diarrhea.
Time Frame: Day 100
Population: 23 patients were able to be analyzed for severe gvhd
Measure: Number; unit: participants
Groups:
- Severe Graft Versus Host Disease: patients receiving transplant using ATG/Bu/Flu/Cy per this protocol and who had severe graft versus host disease as a post-transplant complication
Arm/Group | Severe Graft Versus Host Disease
Number analyzed (Participants) | 23
participants | 2 [0 to 20]

5. Secondary Outcome: Number of Patients Experiencing Extensive Chronic Graft Versus Host Disease (GVHD)
Description: Patients who had post-transplant complication (GVHD) as seen by clinical evidence including but not limited to skin rash, elevated liver function tests, nausea/vomiting/diarrhea.
Time Frame: 2 years
Population: 23 patients were able to be analyzed for severe gvhd
Measure: Number; unit: participants
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Number analyzed (Participants) | 23
participants | 13

6. Secondary Outcome: Non-relapse Mortality (NRM) at Day 180 Post-transplantation
Description: non-relapse mortality refers to the death of a patient for causes other than relapsed disease.
Time Frame: Day 180
Population: 23 patients were able to be analyzed for NRM at 180 days
Measure: Number; unit: participants
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Number analyzed (Participants) | 23
participants | 0

7. Secondary Outcome: Disease-free Survival (DFS) at 24 Months
Description: Disease Free survival is measured by the amount of time a patient spends in a disease free state after being transplanted.
Time Frame: 24 months
Population: 23 patients were able to be analyzed for DFS at 24 months
Measure: Number; unit: participants
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Number analyzed (Participants) | 23
participants | 13 [31 to 72]

8. Secondary Outcome: Overall Survival (OS) at 24 Months
Description: Overall survival refers to the length of time a patient is alive after transplant regardless of whether they have progressive or relapsed disease.
Time Frame: 24 months
Population: 23 patients were able to be analyzed for OS at 24 months
Measure: Number; unit: participants
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Number analyzed (Participants) | 23
participants | 16 [43 to 83]

ADVERSE EVENTS:
Arm/Group | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan
Serious Adverse Events (participants affected / at risk) | 13/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan (N=24)
Abdominal Abcess (Gastrointestinal disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Chemotherapy reaction (General disorders) | 1 (1)
Death (General disorders) | 4 (4)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
GI Bleeding (Gastrointestinal disorders) | 1 (1)
hospitalization for high dose steroid management (General disorders) | 1 (1)
Altered Mental Status (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIC Transplant Using ATG, Busulfan, Fludarabine and Cytoxan (N=24)
abdominal cramping (Gastrointestinal disorders) | 7 (7)
abdominal distension (Gastrointestinal disorders) | 5 (5)
abdominal pain (Gastrointestinal disorders) | 11 (11)
agitation (Social circumstances) | 4 (4)
Alk Phos (Metabolism and nutrition disorders) | 18 (18)
ALT (Metabolism and nutrition disorders) | 17 (17)
altered mental status (Nervous system disorders) | 2 (2)
ANC (Blood and lymphatic system disorders) | 22 (22)
anemia (Blood and lymphatic system disorders) | 21 (21)
anorexia/decreased appetite (Gastrointestinal disorders) | 17 (17)
anxiety (Social circumstances) | 19 (19)
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
AST (Metabolism and nutrition disorders) | 18 (18)
back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
BK virus (Infections and infestations) | 3 (3)
blood in stool (Blood and lymphatic system disorders) | 3 (3)
blurred vision (Eye disorders) | 5 (5)
bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Clostridium difficile (Infections and infestations) | 2 (2)
Chest discomfort (Cardiac disorders) | 2 (2)
chest tightness (Cardiac disorders) | 4 (4)
chest wall pain (Cardiac disorders) | 4 (4)
chills (General disorders) | 17 (17)
CMV (Infections and infestations) | 4 (4)
coarse breath sounds (Respiratory, thoracic and mediastinal disorders) | 2 (2)
confusion (Nervous system disorders) | 4 (4)
constipation (Gastrointestinal disorders) | 9 (9)
cough (Respiratory, thoracic and mediastinal disorders) | 16 (16)
creatinine (Renal and urinary disorders) | 12 (12)
Central venous catheter (CVC) discomfort (Surgical and medical procedures) | 8 (8)
CVC erythema (Skin and subcutaneous tissue disorders) | 2 (2)
dehydration (Metabolism and nutrition disorders) | 3 (3)
depression (Nervous system disorders) | 11 (11)
diaphoresis (Nervous system disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 21 (21)
diminished breath sounds (Respiratory, thoracic and mediastinal disorders) | 2 (2)
dizziness (General disorders) | 9 (9)
drowsy (General disorders) | 7 (7)
dry eye (Eye disorders) | 3 (3)
dry mouth (Gastrointestinal disorders) | 3 (3)
dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
dysphagia (Gastrointestinal disorders) | 6 (6)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (17)
dysuria (Renal and urinary disorders) | 7 (7)
edema (Blood and lymphatic system disorders) | 16 (16)
erythema (Skin and subcutaneous tissue disorders) | 7 (7)
eye irritation (Eye disorders) | 2 (2)
eye redness (Eye disorders) | 2 (2)
Facial flushing (General disorders) | 6 (6)
fall (Musculoskeletal and connective tissue disorders) | 2 (2)
fatigue (General disorders) | 19 (19)
fever (General disorders) | 20 (20)
flat affect (Nervous system disorders) | 3 (3)
flatulence (Gastrointestinal disorders) | 3 (3)
folliculitis (Infections and infestations) | 3 (3)
generalized pain (General disorders) | 7 (7)
Gastroesophogeal Reflux disease (GERD) (Gastrointestinal disorders) | 20 (20)
headache (General disorders) | 21 (21)
hematuria (Renal and urinary disorders) | 2 (2)
hemorrhoids (Gastrointestinal disorders) | 2 (2)
hiccups (General disorders) | 2 (2)
hip pain (Musculoskeletal and connective tissue disorders) | 2 (2)
hyperbilirubinemia (Hepatobiliary disorders) | 10 (10)
hyperglycemia (General disorders) | 20 (20)
hyperkalemia (Metabolism and nutrition disorders) | 18 (18)
hypermagnesemia (Metabolism and nutrition disorders) | 20 (20)
hypernatremia (Metabolism and nutrition disorders) | 5 (5)
hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
hypertension (Cardiac disorders) | 10 (10)
hypoalbuminemia (Metabolism and nutrition disorders) | 23 (23)
hypocalcemia (Metabolism and nutrition disorders) | 19 (19)
hypoglycemia (Metabolism and nutrition disorders) | 5 (5)
hypokalemia (Metabolism and nutrition disorders) | 18 (18)
hypomagnesemia (Metabolism and nutrition disorders) | 20 (20)
hyponatremia (Metabolism and nutrition disorders) | 18 (18)
hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
hypotension (Cardiac disorders) | 4 (4)
hypothyroidism (Endocrine disorders) | 2 (2)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
insomnia (General disorders) | 10 (10)
joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
lethargy (General disorders) | 4 (4)
lip lesion (Skin and subcutaneous tissue disorders) | 2 (2)
lower extremity pain (Musculoskeletal and connective tissue disorders) | 6 (6)
MRSE (Infections and infestations) | 4 (4)
mucositis (Gastrointestinal disorders) | 11 (11)
myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 22 (22)
neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
night sweats (General disorders) | 5 (5)
nocturia (Renal and urinary disorders) | 3 (3)
numbness (Musculoskeletal and connective tissue disorders) | 4 (4)
oral sensitivity (Gastrointestinal disorders) | 7 (7)
Peeling of skin (Skin and subcutaneous tissue disorders) | 2 (2)
petechiae (Blood and lymphatic system disorders) | 3 (3)
pneumonia (Infections and infestations) | 2 (2)
poor appetite (Gastrointestinal disorders) | 3 (3)
post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4)
prurutis (Skin and subcutaneous tissue disorders) | 11 (11)
rash (Skin and subcutaneous tissue disorders) | 11 (11)
restless (General disorders) | 2 (2)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
rigors (General disorders) | 16 (16)
seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 3 (3)
shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8)
skin tenderness (Skin and subcutaneous tissue disorders) | 2 (2)
swelling (hands and fingers) (Blood and lymphatic system disorders) | 2 (2)
tachycradia (Cardiac disorders) | 9 (9)
taste alteration (Gastrointestinal disorders) | 3 (3)
throat pain (Gastrointestinal disorders) | 5 (5)
thrombocytopenia (Blood and lymphatic system disorders) | 23 (23)
thrush (Infections and infestations) | 3 (3)
tremors (Nervous system disorders) | 5 (5)
unsteadiness (Nervous system disorders) | 3 (3)
urinary frequency (Renal and urinary disorders) | 8 (8)
urinary hesitancy (Renal and urinary disorders) | 3 (3)
urinary incontinence (Renal and urinary disorders) | 3 (3)
urinary urgency (Renal and urinary disorders) | 3 (3)
vomiting (Gastrointestinal disorders) | 20 (20)
WBC (leukocytes) (Blood and lymphatic system disorders) | 23 (23)
weakness (General disorders) | 7 (7)
weight gain (General disorders) | 2 (2)
weight loss (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less